CLINICAL TRIAL: NCT05877924
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Anti-tumor Activity of NBL-020 Injection in Subjects With Advanced Malignant Tumors.
Brief Title: A Study of NBL-020 Injection in Subjects With Advanced Malignant Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NovaRock Biotherapeutics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBL-020-001
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-08

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NBL-020 (Experimental): Dose increasing study: The initial dose for the dose escalation study is 0.1 mg/kg administered once every 3 weeks (Q3W), with a pre-set maximum escalation dose of 30 mg/kg Q3W.
  Dose expansion study: Based on the results of the dose escalation study, the dosage for the dose extension study will be determined through joint discussion between the sponsor and the investigators.
  Interventions: Drug: NBL-020 for Injection

INTERVENTIONS:
Drug: NBL-020 for Injection — NBL-020 for Injection, Q3W, i.v.

SUMMARY:
This study aims to evaluate the safety and tolerability of NBL-020 injection in subjects with advanced malignant tumors, and determine the dose limiting toxicity (DLT), maximum tolerable dose (MTD) (if any), recommended phase II dose (RP2D), and dosing regimen of NBL-020.

DETAILED DESCRIPTION:
The study is divided into two parts: dose escalation and dose expansion. Dose increasing study: The initial dose for the dose escalation study is 0.1 mg/kg administered once every 3 weeks (Q3W), with a pre-set maximum escalation dose of 30 mg/kg Q3W. Safety Management Committee (SMC) can jointly discuss and determine whether to proceed with a higher dose group or increase additional doses or different dosing intervals between two adjacent dose groups (such as Q2W or Q4W) based on the safety, tolerance, efficacy, PK, PD, and related biomarker data of each dose group.

Dose expansion study: Based on the results of the dose escalation study, the dosage for the dose extension study will be determined through joint discussion between the sponsor and the investigators. If necessary, multiple doses can be selected for dose extension.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are 18 years old or older (based on the date of signing the informed consent form) and voluntarily sign the informed consent form;
2. For malignant tumors confirmed by histology or cytology, only solid tumor subjects were included in dose escalation study. In addition to solid tumors, additional skin T-cell lymphoma subjects could be considered in dose expansion study;
3. Must be willing to provide tumor tissue samples that can meet the requirements of biomarker testing (fresh biopsy tissue is preferred; if fresh tissue cannot be provided, tumor tissue samples within 2 years can be provided), and tumor samples will be tested by the central laboratory. If tumor tissue does not meet the testing requirements, additional biopsy may be required;
4. If the standard treatment fails or toxicity is intolerable, or there is no standard treatment, the enrolled subjects must fully recover from previous treatment, with an AE level of 0-1 (except for alopecia, pigmentation, or other toxicity that the researcher believes is not a safety risk to the subjects);
5. For subjects with solid tumor, there is at least one measurable lesion that meets the RECIST 1.1 standard at the baseline (the measurable lesion area has not received radiotherapy in the past, or there is evidence that the lesion has unequivocal progressed after radiotherapy);
6. ECOG PS score 0-1 points;
7. Expected survival time ≥ 3 months (12 weeks);
8. Good organ function (no blood transfusion or growth factor support treatment received within 2 weeks before blood collection for relevant examinations), including:

   1. Absolute value of neutrophils (ANC) ≥ 1.5 × 10^9/L；
   2. Hemoglobin (Hb) ≥ 90 g/L;
   3. Platelets ≥ 100 × 10^9 /L;
   4. Creatinine ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance rate ≥ 50 mL/min (Cockcroft Fault formula);
   5. Total bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for Gilbert's syndrome）;
   6. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for subjects with liver metastasis);
   7. Coagulation function: activated partial thromboplastin time(APTT), international standardized ratio (INR) ≤ 1.5 × ULN.

   Note: If the subject does not meet the requirements during screening, a re-examination is allowed.
9. The subjects must agree to take effective contraceptive measures from the signing of the informed consent form until 6 months after the last administration. Women of childbearing age tested negative for serum pregnancy within 7 days before the first dose of the investigational drug.

Exclusion Criteria:

1. Subjects with a history of severe allergies to monoclonal antibodies;
2. Active pia mater lesions or uncontrolled brain metastases exist. Subjects with suspected or confirmed brain metastasis can be enrolled as long as they are asymptomatic and do not require treatment (such as radiotherapy, surgery, or corticosteroid therapy) to control the symptoms of brain metastasis. For subjects with brain metastasis requiring treatment, their symptoms remain stable (without hormone maintenance treatment, without symptoms of brain metastasis) for 2 weeks after treatment, and they can be enrolled.
3. Subjects with active autoimmune diseases or a history of autoimmune diseases, but with the following diseases are allowed to be included in the study: well controlled type I diabetes, well controlled hypothyroidism only requiring hormone replacement treatment, skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia), or subjects who are expected to have no relapse under the condition of no external trigger factors;
4. Having a history of primary immunodeficiency, a history of allogeneic organ transplantation, or a history of allogeneic hematopoietic stem cell transplantation;
5. Chronic hepatitis B (HBsAg and/or HBcAb positive but HBV DNA<2000 IU/mL can be included), chronic hepatitis C (HCV antibody positive but HCV RNA negative can be included), and HIV antibody positive;
6. The toxicity of previous anti-tumor treatments has not returned to ≤ Grade 1 (except for alopecia, pigmentation, or other toxicity that the researchers believe is not a safety risk to the subjects);
7. Have a history of serious cardiovascular disease, including but not limited to:

   1. Serious cardiac rhythm or conduction abnormalities, including but not limited to ventricular arrhythmias requiring clinical intervention, third degree atrioventricular block, within 6 months prior to the first dose of the investigational drug;
   2. Have a history of myocardial infarction, unstable angina, angioplasty, or coronary artery bypass surgery within 6 months before the first dose of the experimental drug;
   3. Heart failure, classified as Grade Ш or above by the New York Heart Association (NYHA);
   4. Subjects with prolonged QT/QTc interval in the screening period electrocardiogram);
   5. During the screening, echocardiography showed left ventricular ejection fraction (LVEF)<50%;
   6. Poor control of hypertension (screening period systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
8. Uncontrollable serous cavity effusion that requires frequent drainage or medical intervention (such as pleural effusion, abdominal effusion, pericardial effusion, etc., which requires additional intervention within 2 weeks after the intervention, excluding exfoliative cytology testing of the exudate) within 7 days before the first dose of the experimental drug;
9. Severe or active infections (including tuberculosis infections) that require systemic antibacterial, antifungal, or antiviral treatment within 14 days before the first use of the experimental drug, except for subjects with viral hepatitis receiving antiviral treatment;
10. Received any anti-tumor treatment (including chemotherapy, targeted therapy, immunotherapy, etc.) and any clinical research treatment within 4 weeks or 5 half-lives before the first administration (whichever is shorter);
11. Have a history of (non-infectious) pneumonia/interstitial lung disease requiring steroid treatment, or currently have (non-infectious) pneumonia/interstitial lung disease requiring steroid treatment.
12. Subjects are required to receive systemic corticosteroids (>10 mg daily prednisone or equivalent) or immunosuppressive therapy within 14 days before the first dose. Inhalation or local application of corticosteroids, adrenal hormone replacement therapy, and short-term (≤ 7 days) use of corticosteroids to prevent contrast agent allergies are allowed.
13. History of immune related adverse events (immune-related AE) ≥ Grade 3 (CTCAE 5.0) after receiving immunotherapy;
14. Previously received targeted TNFR2 treatment;
15. Those who have undergone major surgery within 4 weeks before the first administration and have not yet fully recovered, or plan to undergo major surgery during the study period;
16. Previous malignancies other than the disease under study within 3 years, except for those that can be cured through local treatment, such as skin basal cell carcinoma, cervical or breast cancer in situ;
17. Pregnant or lactating women;
18. Participate in another clinical study at the same time, unless it is an observational (non-intervention) clinical study or during the follow-up period of an intervention study;
19. Has a clear history of neurological or mental disorders, including epilepsy or dementia;
20. Other circumstances that researchers believe not suitable to participate in clinical trials, including but not limited to: subjects with severe or uncontrollable medical conditions, safety risks, interference with the interpretation of research results, and impact on trial compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of all adverse events (AEs) and severe adverse events (SAEs). | From the first administration to 30 days after the end of the last administration, up to approximately 2 years
  adverse events (AEs) and severe adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax | 14 days
  Observed maximum concentration
AUC0-t | 14 days
  AUC0-t
AUC0-inf | 14 days
  AUC0-inf
Tmax | 14 days
  Time to maximum concentration
t1/2 | 14 days
  Apparent terminal Half-Life
Vz | 14 days
  Vz
ORR | Up to approximately 2 years.
  Objective response rate
DCR | Up to approximately 2 years.
  Disease control rate
PFS | Up to approximately 2 years.
  Progression free survival
DOR | Up to approximately 2 years.
  Duration of response
OS | Up to approximately 2 years.
  Overall survival
Anti NBL-020 antibody (ADA) and neutralizing antibody (Nab). | 14 days
  Anti NBL-020 antibody and neutralizing antibody.
NBL-020 receptor occupancy rate for tumor necrosis factor type Ⅱ receptor (TNFR2). | 14 days
  NBL-020 receptor occupancy rate for tumor necrosis factor type Ⅱ receptor.
Concentration of free tumor necrosis factor type Ⅱ receptor (TNFR2). | 14 days
  Concentration of free tumor necrosis factor type Ⅱ receptor.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital, Guangzhou City, Guangdong Province, China
Locations (1):
- Wu Yilong, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No